CLINICAL TRIAL: NCT06550713
Title: Phase I Clinical Trial Protocol for Tolerability and Pharmacokinetics of TQB3455 Tablets in Patients With Hematological Malignancies
Brief Title: A Clinical Trial of TQB3455 Tablets in Patients With Hematological Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3455-I-01
Record Dates: First submitted 2022-07-25; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Acute Myeloid Leukemia (AML); Myelodysplastic Syndrome (MDS)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3455 tablet and Azacitidine for Injection (Experimental): Stage1：TQB3455 tablet, oral, once a day, for 28 consecutive days as a treatment cycle.
  Stage2：TQB3455 tablet, oral, once a day, for 28 consecutive days as a treatment cycle.
  Azacitidine for injection: A treatment cycle of 4 weeks, with subcutaneous injection of Azacitidine standard dose on the first to seventh day of each cycle.
  Interventions: Drug: TQB3455 tablet+Azacitidine for Injection

INTERVENTIONS:
Drug: TQB3455 tablet+Azacitidine for Injection — TQB3455 is a selective IDH2 mutant enzyme inhibitor. Azacitidine for injection is a cytosine nucleoside drug that is used for demethylation therapy.

SUMMARY:
This study is a clinical trial to evaluate the tolerability and pharmacokinetics of TQB3455 tablets in patients with hematological malignancies. TQB3455 is an isocitrate dehydrogenase 2(IDH2) inhibitor . This project is divided into two stages. The first stage aims to evaluate the safety and tolerability of single or multiple oral administration of TQB3455 tablets in subjects with malignant hematological tumors. The second phase aims to evaluate the efficacy and safety of TQB3455 tablets alone or in combination with azacitidine in subjects with acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS).

ELIGIBILITY:
Inclusion Criteria:

Patients meeting all of the following inclusion criteria can be included in this trial:

* Age ≥ 18 years old;
* According to the World Health Organization (WHO) classification, subjects diagnosed with myelodysplastic syndrome (MDS) and acute myeloid leukemia (AML) should meet one of the following criteria:

  1. Difficult to treat or recurrent (>5% of primitive cells reappear in the bone marrow after complete remission) AML; (Single drug group)
  2. Newly diagnosed AML subjects recognized by researchers as unable to receive standard treatment due to age, physical condition, or risk factors; (Joint group)
* MDS subjects belong to the following prognostic risk categories according to the revised International Prognostic Scoring System (IPSS-R):

  1. Extremely high-risk (>6 points)
  2. High risk (>4.5 points - ≤ 6 points)
  3. Medium risk (>3 points - ≤ 4.5 points)
* Clearly indicating the presence of IDH2 gene mutation;
* Blood platelet (PLT) ≥20×10^9/L； Or subjects with PLT<20 × 10^9/L, but recognized by the researchers as being caused by tumor reasons;
* Serum total bilirubin ≤ 1.5 × ULN (for Gilbert syndrome subjects, bilirubin ≤ 3 × ULN);
* Renal function: serum creatinine ≤ 1.5 × ULN or creatinine clearance rate ≥ 50ml/min;
* Recovery of toxic reactions caused by surgery, radiation therapy, or other anti-tumor treatments to ≤ Grade I;
* Women should agree to use contraceptive measures during the study period and within 6 months after the end of the study; Male participants must agree to use contraception during the study period and within 6 months after the end of the study period;
* The subjects voluntarily joined this study.

Exclusion Criteria:

* Subjects who experience relapse after bone marrow transplantation;
* Subjects who have received systemic anti-tumor therapy or radiation therapy within 3 weeks prior to the use of the investigational drug;
* Individuals who have participated in clinical trials of other drugs within the four weeks prior to using the investigational drug;
* Individuals with multiple factors that affect oral medication, such as inability to swallow, post gastrointestinal resection, chronic diarrhea, and intestinal obstruction;
* Subjects who have previously used targeted isocitrate dehydrogenase 2 (IDH2) inhibitors;
* The subject has uncontrolled systemic fungal, bacterial, or viral infections;
* High blood pressure subjects who are still poorly controlled despite drug treatment;
* Obvious cardiovascular diseases, such as heart failure classified as grade 2 or above by the New York Heart Association (NYHA), unstable angina in the past 3 months, myocardial ischemia or infarction, arrhythmia and grade I heart failure, or the presence of other factors at risk of prolonging the QT interval (such as arrhythmia, hypokalemia ≥ grade 3, family history of long QT interval);
* Severe leukemia complications that endanger life, such as uncontrolled bleeding, hypoxia or shock pneumonia, disseminated intravascular coagulation;
* Subjects known to have central nervous system leukemia or clinical symptoms of central nervous system leukemia;
* Individuals with a history of abuse of psychotropic drugs who are unable to quit or have mental disorders;
* Subjects with active replication of hepatitis B virus and hepatitis C virus;
* Individuals with a history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
* According to the researcher's judgment, there are accompanying diseases that pose a serious threat to the safety of the subjects or affect their ability to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-10-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Baseline up to 28 days
  Subjects appear the toxic reaction relate to the drug after treatment within 28 days.
The maximum tolerated dose (MTD) | Up to 48 weeks
  The highest dose at which no more than 33% of the subjects experience a dose-limiting toxicity (DLT) during treatment.
Overall Remission Rate | Up to 48 weeks
  The number of participants with CR + incomplete recovery (CRi) + incomplete platelet recovery (CRp) according to modified International Working Group Acute Myeloid Leukemia (IWG AML) response criteria.

SECONDARY OUTCOMES:
Overall survival (OS) | U to 96 weeks
  Overall survival defined as the time from enrollment to death from any cause.
Duration of Response (DOR) | Up to 48 weeks
  DOR will be defined as median number of months from date of first documented objective response until first documented sign of disease progression or death due to any causes.
Complete Remission Rate | Up to 48 weeks
  The number of participants with morphologic complete remission (CR) according to modified International Working Group Acute Myeloid Leukemia Response Criteria (IWG AML).
Cmax | Hour 0, 0.25, 0.5, 1, 2, 3, 5, 8, 10, 12, 24, 48, 96, 144 hours post-dose on single dose; Hour 0 of day 8, day 15, day 22 on multiple dose and hour 0, 0.25, 0.5, 1, 2, 3, 5, 8, 12, 24 hours post-dose on multiple dose of day 28
  Cmax is the maximum plasma concentration of TQB3455 or metabolite(s).
Tmax | Hour 0, 0.25, 0.5, 1, 2, 3, 5, 8, 10, 12, 24, 48, 96, 144 hours post-dose on single dose; Hour 0 of day 8, day 15, day 22 on multiple dose and hour 0, 0.25, 0.5, 1, 2, 3, 5, 8, 12, 24 hours post-dose on multiple dose of day 28
  To characterize the pharmacokinetics of TQB3455 by assessment of time to reach maximum plasma concentration.
Area Under the Curve (AUC) 0-t | Hour 0, 0.25, 0.5, 1, 2, 3, 5, 8, 10, 12, 24, 48, 96, 144 hours post-dose on single dose; Hour 0 of day 8, day 15, day 22 on multiple dose and hour 0,0.25, 0.5, 1, 2, 3, 5, 8, 12, 24 hours post-dose on multiple dose of day 28
  To characterize the pharmacokinetics of TQB3455 by assessment of area under the plasma concentration time curve from zero to infinity.
α-Hydroxyglutaric acid (2-HG) | Day 1, Day 8 and Day 15 pre-dose on cycle 1; Day1, Day15 pre-dose on cycle 2 ; Day 1 pre-dose on multiple dose from cycle 3 to cycle 8. Each cycle is 28 days.
  The concentration of 2-HG.

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Peking University international Hospital, Beijing, Beijing Municipality
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin The First Hospital, Harbin, Heilongjiang
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - People's Hospital of Tianjin, Tianjin, Tianjin Municipality